CLINICAL TRIAL: NCT06702735
Title: The Rainbow Study - a Randomized Controlled Trial to Evaluate the Effect of Personalized Feedback on Symptom Perception in Asthmatic Children
Brief Title: The Rainbow Study - the Effect of Feedback on Asthmatic Symptom Perception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RAINBOW study
Record Dates: First submitted 2023-10-16; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Asthma in Children; Exercise Induced Asthma
MeSH Terms: conditions — Asthma, Exercise-Induced

STUDY DESIGN:
Intervention Model Description: This study is a prospective, non-blinded randomized controlled trial with three parallel arms. After a selection phase of 2 weeks, eligible participants were equally allocated to the study arms (ratio 1:1:1). The intervention phase consists of three weeks, followed by a follow-up of two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group (with feedback) (Experimental): Collection of VAS scores and lung function. Explanation about the Rainbow tool to visualize symptom perception, and use of this tool during intervention phase. Feedback sessions with health care professional to evaluate symptom perception using the Rainbow tool.
  Interventions: Behavioral: Rainbow tool; Behavioral: Feedback
- Intervention group (without feedback) (Experimental): Collection of VAS scores and lung function. Explanation about the Rainbow tool to visualize symptom perception, and use of this tool during intervention phase.
  Interventions: Behavioral: Rainbow tool
- Control group (No Intervention): Collection of VAS scores and lung function. No additional intervention.

INTERVENTIONS:
Behavioral: Rainbow tool — The Rainbow tool visualizes perception based on lung function measurements and VAS scores.
  Arms: Intervention group (with feedback); Intervention group (without feedback)
Behavioral: Feedback — Feedback sessions with health care professional based on the Rainbow tool.
  Arms: Intervention group (with feedback)

SUMMARY:
Asthma is a common childhood disease that is characterized by chronic airway inflammation and episodic expiratory airflow obstruction. Asthma symptoms can impair participation in play and sports and have a negative impact on quality of life. It can be challenging for children to adequately feel and report their symptoms. Some children experience more symptoms than expected based on lung function during these symptoms, whereas others experience less symptoms than expected. This is also called 'symptom perception'.

A tool was developed to visualize symptoms, lung function and accessory symptom perception: The Rainbow tool. The aim of this study was to identify asthmatic children with a poor perception and investigate if their symptom perception could be improved by regular lung function measurements and personal feedback based on the Rainbow Tool.

Hypothesis: Measuring lung function en symptoms and provide personal feedback on perception based on the Rainbow tool has a positive effect on perception of asthma-related symptoms in asthmatic children.

DETAILED DESCRIPTION:
Asthma is a common childhood disease that is characterized by chronic airway inflammation and episodic expiratory airflow obstruction. Asthma symptoms can impair participation in play and sports and have a negative impact on quality of life. It can be challenging for children to adequately feel and report their symptoms. Some children experience more symptoms than expected based on lung function during these symptoms, whereas others experience less symptoms than expected. This is also called 'symptom perception'.

A tool was developed to visualize symptoms, lung function and accessory symptom perception: The Rainbow tool. The Rainbow tool is a two-dimensional color-coded plot, visualizing the relationship between lung function, denoted as a percentage of personal best (FEV1) on the vertical axis, and VAS score on the horizontal axis. The FEV1 as a percentage of personal best on the vertical axis ranges from 30% to 100% since a maximal VAS score would be expected with a change in FEV1 to ≤ 30% of personal best. The horizontal axis ranges from 0 to 10, with 0 indicating no dyspnea and 10 maximal dyspnea. There are four color-coded zones: the green zone, yellow zone, orange zone, and red zone. The green zone indicates good alignment between symptoms and lung function, and thus a good symptom perception. It forms a diagonal band from the upper left (around 100% FEV1 and VAS score of 0) stretching to the lower right (around 30% FEV1 and VAS score of 10). The green zone is followed by the yellow, orange, and red zones on either side, indicating an increasing deviation in symptom perception from the ideal and respectively mild, moderate, and severe disconcordance between FEV1 and VAS score. The aim of this study was to identify asthmatic children with a poor perception and investigate if their symptom perception could be improved by regular lung function measurements and personal feedback based on the Rainbow Tool.

Hypothesis: Measuring lung function en symptoms and provide personal feedback on perception based on the Rainbow tool has a positive effect on perception of asthma-related symptoms in asthmatic children.

ELIGIBILITY:
Inclusion Criteria:

Selection phase:

* Pediatrician diagnosed asthma
* Health care professional thinks perception might be poor
* Age 7 until 15 years old
* Adequate understanding of Dutch language

Intervention phase:

* Adequate number of lung function measurements + VAS scores during selection phase, defined as:
* At least 4 measurements after exercise or when experiencing symptoms and
* At least 2 standard measurements
* Poor perception during selection phase, defined as:
* At least 1 measurement in red zone on Perception Rainbow and/or
* At least 2 measurements in orange zone on Perception Rainbow and/or
* Average of all measurements after exercise or when experiencing symptoms in yellow zone (or orange/red)and/or
* Average of all measurements in yellow zone (or orange/red)

Exclusion Criteria:

* Severe comorbidity (for example psychomotor retardation or severe cardiopulmonary conditions)
* Not able to fill in VAS score (for example due to blindness)
* Not able to perform technically correct spirometry manoeuvres
* Medication change in past 2 weeks
* Exacerbation which required oral prednisone in the past 6 weeks
* Exacerbation at the moment of inclusion
* No device (computer, tablet or smartphone) with internet connection available at home

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Perception score | Two week run-in versus last week of intervention
  The difference in the average perception score (0-100) during the two-week run-in and last week of the intervention between the intervention group (with feedback) and the control group

SECONDARY OUTCOMES:
Perception score intervention groups | Measured per week during the study period, which is 8 weeks
  Difference between average perception score of intervention group (with feedback) and intervention (without feedback) group per week
Perception score over time | Measured per week during the study period, which is 8 weeks
  Perception scores (0-100) and average perception score per week. Including over- or underperception
Perception score zones | Measured per week during the study period, which is 8 weeks
  Number of perception scores in green/yellow/red zone (absolute and relative) per week
Additional symptoms | Measured per week during the study period, which is 8 weeks
  Type of additional symptom when measurement (lung function + VAS) is performed: no additional symptoms, cough, wheezing, chest pain, feeling dizzy, nasal symptoms
Drop-out rate | Per study phase, 2 weeks for selection phase, 3 weeks for intervention phase and 3 weeks for follow-up phase
  Number of patients that drop-out during or after selection phase and reasons for drop-out
User experience | After the intervention phase, that takes 3 weeks
  User experience based on semi-structured interview and user experience + technology acceptance questionnaire after the intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Vera Hengeveld, MD, Principal Investigator — Medisch Spectrum Twente
Locations (1):
- Medisch Spectrum Twente, Enschede, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No